CLINICAL TRIAL: NCT04621682
Title: Non-technical Skills Training and Checklists Versus Standard Training With Checklists in Boarding School Students to Reduce Simulation Crisis Medical Error, Randomized Controlled Clinical Trial
Brief Title: Non-technical Skills Training and Checklists Versus Standard Training With Checklists for Prevention of Medical Error
Acronym: TECRISIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Mario Zamudio, Clinical Professor, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: F070
Record Dates: First submitted 2020-06-12; First posted 2020-11-09 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Medical Emergencies
Keywords: medical error; high fidelity simulation; non technical skills; checklist

STUDY DESIGN:
Intervention Model Description: TECRISIS is a study designed as a controlled clinical trial of superiority with parallel groups, random allocation and blinding of investigators who measure outcome.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non technical skills and check list (Active Comparator): 10 hours of training in non-technical skills and checklists in high Fidelity simulation
  Interventions: Other: Non technical skills and checklist training in simulation
- check list (Active Comparator): Control: 10 hours of standard training with checklists in high Fidelity simulation
  Interventions: Other: Checklist training simulation

INTERVENTIONS:
Other: Non technical skills and checklist training in simulation — using structured debrifing, in three random medical simulation crises, training in non-technical skills will be carried out
  Arms: Non technical skills and check list
Other: Checklist training simulation — using structured debrifing, in three random medical simulation crises, training in checklist will be carried out
  Arms: check list

SUMMARY:
The purpose of this study is to reduce medical error by omitting management steps in medical crises. The Interventions will be: training in non-technical skills and checklists versus Control: standard training with checklists

DETAILED DESCRIPTION:
56 participants will be searched for simulation training, randomly assigned in assignment 1 to 1, the follow-up will be 10 days, the primary outcome will be Proportion of omissions of treatment steps per group, and secondary outcomes will be sought. Crisis resolution time, detection time. and discrimination from the crisis Global score of non-technical skills, Discriminated score between dimensions of non-technical skills, Student satisfaction and Incidence of inadequate crisis management.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old.
* Final semester student of medicine at the University of Antioquia.
* Have passed the theoretical knowledge exam for handling crisis events with a score of 100%.
* On-site availability on training days

Exclusion Criteria:

* Having received training in a specific crisis resource management course.
* Refusing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-07-18 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Medical error | 3 days after finishing the training
  Proportion of omission of treatment steps over the total number of steps per group.

SECONDARY OUTCOMES:
Overall score on non-technical skills scale Ottawa | 3 days after finishing the training
  Mean interval difference per group between 1 to 45
  Brief Name: Ottawa Global Rating Scale (GRS) Minimum value: 1 Maximum value: 45 Higher scores mean a better outcome
score for each non-technical skill category on the ottawa scale | 3 days after finishing the training
  Mean interval difference per group between 1 to 7
  Brief Name: Ottawa Global Rating Scale (GRS)/ For Category Minimum value: 1 Maximum value: 7 Higher scores mean a better outcome
Crisis resolution time | 3 days after finishing the training
  Mean interval difference per group
Time in detection and discrimination of the crisis | 3 days after finishing the training
  Mean interval difference per group
Incidence of improper handling | 3 days after finishing the training
  relative risk
Student understanding of strategies | 10 days after finishig the primary outcome
  qualitative analysis with grounded theory after conducting semi-structured interviews

CONTACTS AND LOCATIONS:
Locations (1):
- Mario Andres Zamudio, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: Yes
through email communication with the lead author
Supporting Information: Study Protocol
Time Frame: 10 years
Access Criteria: through email communication with the lead author

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/82/NCT04621682/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/82/NCT04621682/ICF_001.pdf